CLINICAL TRIAL: NCT04853238
Title: COPD Disease Burden, Patient Characteristics, Maintenance Treatment Patterns and Factors Influencing Treatment Decisions in China Tier 2 and Tier 3 Hospitals
Brief Title: Chronic Obstructive Pulmonary Disease (COPD) Maintenance Treatment Patterns in China
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 213550
Record Dates: First submitted 2021-04-16; First posted 2021-04-21 (Actual); Results first posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Chronic obstructive pulmonary disease; China; Disease burden; Maintenance treatment patterns
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort 1: Participants with stable disease
  Interventions: Other: Prospective observational cohort study
- Cohort 2: Participants with moderate acute exacerbation not requiring hospitalization
  Interventions: Other: Prospective observational cohort study
- Cohort 3: Participants requiring hospitalization for an acute exacerbation
  Interventions: Other: Prospective observational cohort study

INTERVENTIONS:
Other: Prospective observational cohort study — Prospective observational cohort study. No study treatment was administered in this study.

SUMMARY:
This observational study will be conducted in COPD participants in Tier 2 and 3 hospitals in China to gain an understanding of the complex COPD management and physician's treatment strategy.

ELIGIBILITY:
Inclusion criteria:

* Male or female participants with minimum 40 years of age.
* A diagnosis of COPD confirmed by spirometry (According to Global initiative for chronic obstructive lung disease [GOLD] 2019 criteria) in Tier 2 and Tier 3 hospitals.
* In hospitalized participants, recruit only participants who receive any intravenous therapy.
* A signed and dated written informed consent.
* Participants can communicate normally.

Exclusion criteria:

* Current primary diagnosis of asthma, active tuberculosis, bronchiectasis, lung cancer or other active pulmonary disease.
* Other unstable diseases or cognitive behavior, which could influence CAT and lung function results (judged by physicians).
* Experienced a moderate/severe COPD exacerbation treated by a physician within last 1 month.
* Currently participating in another COPD clinical study, which provides the participant investigational medication and/or disease management.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with COPD either in stable state or with an acute exacerbation, in Tier 2 and 3 hospitals in China.
Sampling Method: Non-Probability Sample
Enrollment: 1507 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2022-11-03 (Actual); Study Completion 2023-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (33):
- China (33):
  - GSK Investigational Site, Huizhou, Guangdong
  - GSK Investigational Site, Jiangmen, Guangdong
  - GSK Investigational Site, Shaoguan, Guangdong
  - GSK Investigational Site, Shenzhen, Guangdong
  - GSK Investigational Site, Nanning, Guangxi
  - GSK Investigational Site, Wuhan, Hubei
  - GSK Investigational Site, Shenyang, Liaoning
  - GSK Investigational Site, Yinchuan, Ningxia
  - GSK Investigational Site, Xi'an, Shaanxi
  - GSK Investigational Site, Jinan, Shandong
  - GSK Investigational Site, Taiyuan, Shanxi
  - GSK Investigational Site, Zhejiang, Zhejiang
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Cangzhou
  - GSK Investigational Site, Chengdu
  - GSK Investigational Site, Chongqing
  - GSK Investigational Site, Hangzhou
  - GSK Investigational Site, Hefei
  - GSK Investigational Site, Jingzhou
  - GSK Investigational Site, Luoyang
  - GSK Investigational Site, Nanchang
  - GSK Investigational Site, Nanning
  - GSK Investigational Site, Nanyang
  - GSK Investigational Site, Pingdingshan
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Shanxi
  - GSK Investigational Site, Shenyang
  - GSK Investigational Site, Tianjin
  - GSK Investigational Site, Wuhan
  - GSK Investigational Site, Xi'an
  - GSK Investigational Site, Xiangtan
  - GSK Investigational Site, Yibin
  - GSK Investigational Site, Zhengzhou

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This non-interventional study aims to assess Chronic Obstructive Pulmonary Disease (COPD) maintenance treatment patterns among newly diagnosed and previously diagnosed participants with COPD presenting to clinics, either in a stable state or with acute exacerbation. No study treatment was administered in current study (NCT04853238).
Pre-assignment Details: A total of 1507 participants were enrolled in the study (Enrolled Population: All participants who passed screening [met eligibility criteria] and entered the study).
Groups:
- Cohort 1: Participants Presenting With Stable Disease: Participants with newly diagnosed and previously diagnosed COPD presenting to clinics in a stable state (no exacerbation for at least 1 month) were included in this cohort.
- Cohort 2: Participants Presenting With a Moderate Acute Exacerbation Not Requiring Hospitalization: Participants with newly diagnosed and previously diagnosed COPD with moderate acute exacerbations not requiring hospitalization were included in this cohort.
- Cohort 3: Participants Requiring Hospitalization for an Acute Exacerbation: Participants with newly diagnosed and previously diagnosed COPD with acute exacerbation requiring hospitalization were included in this cohort.
Period: Overall Study
Arm/Group | Cohort 1: Participants Presenting With Stable Disease | Cohort 2: Participants Presenting With a Moderate Acute Exacerbation Not Requiring Hospitalization | Cohort 3: Participants Requiring Hospitalization for an Acute Exacerbation
Started (Enrolled) | 802 | 71 | 634
Analysis Data Set | 797 | 71 | 615
Completed | 772 | 68 | 561
Not Completed | 30 | 3 | 73
Not completed — Death | 4 | 0 | 2
Not completed — Lost to Follow-up | 16 | 2 | 37
Not completed — Poor adherence, unable to cooperate with investigator to complete test | 1 | 1 | 10
Not completed — Withdrawal by Subject | 6 | 0 | 21
Not completed — Physician Decision | 0 | 0 | 2
Not completed — Violation of inclusion/exclusion criteria | 3 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline Characteristic data are reported for Analysis data set which included all participants from enrolled population excluding those who did not enter the study as they did not meet Protocol-defined eligibility criteria.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Participants Presenting With Stable Disease | Cohort 2: Participants Presenting With a Moderate Acute Exacerbation Not Requiring Hospitalization | Cohort 3: Participants Requiring Hospitalization for an Acute Exacerbation | Total
Number analyzed (Participants) | 797 | 71 | 615 | 1483
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.1 (8.15) | 68.3 (8.40) | 69.1 (8.28) | 68.0 (8.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 5 | 69 | 168
  Male | 703 | 66 | 546 | 1315
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian-Chinese | 797 | 71 | 615 | 1483

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Received COPD Prescription for Maintenance Treatment at Baseline
Description: Participants who received prescription for COPD maintenance treatment were reported for following categories; Use the maintenance treatment, Long-Acting Muscarinic Antagonist (LAMA), Long-Acting Beta-Agonist (LABA), LABA/LAMA, inhaled corticosteroid (ICS)/LABA, Triple therapy (ICS/LABA/LAMA, Single Inhaler Triple Therapy [SITT]), Multiple Inhaler Triple Therapy (MITT), Theophylline, MITT or SITT, N-acetyl cysteine/carbocysteine. The measurement at Baseline visit (Day 1) was defined as Baseline. Participants may have received more than one COPD maintenance treatment. Hence, they may have counted in more than one category, so the total may not match to Number analyzed (N).
Time Frame: At Baseline (Day 1)
Population: Analysis data set which included all participants from enrolled population excluding those who did not enter the study as they did not meet Protocol-defined eligibility criteria. Only those participants who were measured and analyzed (i.e., contributed data reported in the table) were included in the 'Overall Number of Participants Analyzed' field.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Participants Presenting With Stable Disease | Cohort 2: Participants Presenting With a Moderate Acute Exacerbation Not Requiring Hospitalization | Cohort 3: Participants Requiring Hospitalization for an Acute Exacerbation
Number analyzed (Participants) | 797 | 71 | 615
Participants
  Use the maintenance treatment | 735 | 68 | 554
  LAMA | 105 | 3 | 13
  LABA | 1 | 0 | 0
  LABA/LAMA | 164 | 16 | 34
  ICS/LABA | 165 | 20 | 107
  Triple therapy (ICS/LABA/LAMA, SITT) | 225 | 17 | 126
  MITT | 55 | 6 | 43
  Theophylline | 117 | 12 | 427
  MITT or SITT | 280 | 23 | 169
  N-acetyl cysteine/carbocysteine | 81 | 16 | 240

2. Primary Outcome: Number of Participants Who Received COPD Prescription for Maintenance Treatment at 3 Months
Description: Participants who received prescription for COPD maintenance treatment were reported for following categories; Use the maintenance treatment, LAMA, LABA, LABA/LAMA, ICS/LABA, Triple therapy (ICS/LABA/LAMA, SITT), MITT, Theophylline, MITT or SITT, N-acetyl cysteine/carbocysteine. Participants may have received more than one COPD maintenance treatment. Hence, they may have counted in more than one category, so the total may not match to Number analyzed (N).
Time Frame: At 3 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Participants Presenting With Stable Disease | Cohort 2: Participants Presenting With a Moderate Acute Exacerbation Not Requiring Hospitalization | Cohort 3: Participants Requiring Hospitalization for an Acute Exacerbation
Number analyzed (Participants) | 797 | 71 | 615
Participants
  Use the maintenance treatment | 685 | 57 | 433
  LAMA | 95 | 6 | 26
  LABA | 1 | 0 | 0
  LABA/LAMA | 138 | 12 | 36
  ICS/LABA | 143 | 20 | 115
  Triple therapy (ICS/LABA/LAMA, SITT) | 241 | 13 | 186
  MITT | 46 | 3 | 41
  Theophylline | 91 | 7 | 80
  MITT or SITT | 287 | 16 | 227
  N-acetyl cysteine/carbocysteine | 69 | 9 | 57

3. Primary Outcome: Number of Participants With Moderate Acute Exacerbation Requiring no Hospitalization by Each COPD Maintenance Treatment at Follow-up (Week 1)
Description: Participants with moderate acute exacerbation requiring no hospitalization, who received prescription for COPD maintenance treatment were reported for following categories; Use the maintenance treatment, LAMA, LABA, LABA/LAMA, ICS/LABA, Triple therapy (ICS/LABA/LAMA, SITT), MITT, Theophylline, MITT or SITT, N-acetyl cysteine/carbocysteine. Participants may have received more than one COPD maintenance treatment. Hence, they may have counted in more than one category, so the total may not match to Number analyzed (N).
Time Frame: At Week 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: Participants Presenting With a Moderate Acute Exacerbation Not Requiring Hospitalization
Number analyzed (Participants) | 71
Participants
  Use the maintenance treatment | 17
  LAMA | 3
  LABA | 0
  LABA/LAMA | 1
  ICS/LABA | 3
  Triple therapy (ICS/LABA/LAMA, SITT) | 2
  MITT | 0
  Theophylline | 5
  MITT or SITT | 2
  N-acetyl cysteine/carbocysteine | 6

4. Primary Outcome: Number of Participants With Acute Exacerbation Requiring Hospitalization by Each COPD Maintenance Treatment at Discharge Follow-up (up to 28 Days)
Description: Participants with acute exacerbation requiring hospitalization who received prescription for COPD maintenance treatment were reported for following categories; Use the maintenance treatment. LAMA, LABA, LABA/LAMA, ICS/LABA, Triple therapy (ICS/LABA/LAMA, SITT), MITT, Theophylline, MITT or SITT, N-acetyl cysteine/carbocysteine. Participants may have received more than one COPD maintenance treatment. Hence, they may have counted in more than one category, so the total may not match to Number analyzed (N).
Time Frame: At Discharge follow-up (up to 28 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Participants Requiring Hospitalization for an Acute Exacerbation
Number analyzed (Participants) | 615
Participants
  Use the maintenance treatment | 537
  LAMA | 29
  LABA | 0
  LABA/LAMA | 63
  ICS/LABA | 131
  Triple therapy (ICS/LABA/LAMA, SITT) | 196
  MITT | 51
  Theophylline | 164
  MITT or SITT | 247
  N-acetyl cysteine/carbocysteine | 157

5. Secondary Outcome: Mean Forced Expiratory Volume in One Minute (FEV1) at Baseline
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one minute. FEV1 measurements were collected using a spirometer. The measurement at Baseline visit (Day 1) was defined as Baseline.
Time Frame: At Baseline (Day 1)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Cohort 1: Participants Presenting With Stable Disease | Cohort 2: Participants Presenting With a Moderate Acute Exacerbation Not Requiring Hospitalization | Cohort 3: Participants Requiring Hospitalization for an Acute Exacerbation
Number analyzed (Participants) | 797 | 71 | 600
Liters | 1.424 (0.6313) | 1.405 (0.6178) | 1.137 (0.5312)

6. Secondary Outcome: Number of Participants With History of Exacerbations in Within 1 Year Prior to Baseline
Description: Number of participants with history of exacerbations were reported according to the usage of different patterns of maintenance therapy including LAMA, LABA, LABA/LAMA, ICS/LABA, Triple therapy (ICS/LABA/LAMA, SITT), MITT, Theophylline, MITT or SITT, N-acetyl cysteine/carbocysteine. The measurement at Baseline visit (Day 1) was defined as Baseline. Participants may have received more than one COPD maintenance treatment. Hence, they may have counted in more than one category, so the total may not match to Number analyzed (N).
Time Frame: Within 1 year prior to Baseline (Day 1) visit
Population: Analysis data set which included all participants from enrolled population excluding those who did not enter the study as they did not meet Protocol-defined eligibility criteria. All participants who were measured and analyzed (i.e., contributed data reported in the table) were included in the 'Overall Number of Participants Analyzed' field. 'Number Analyzed' signifies participants evaluable for the specified time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Participants Presenting With Stable Disease | Cohort 2: Participants Presenting With a Moderate Acute Exacerbation Not Requiring Hospitalization | Cohort 3: Participants Requiring Hospitalization for an Acute Exacerbation
Number analyzed (Participants) | 797 | 71 | 615
Participants
  LAMA: number analyzed (Participants) | 75 | 0 | 15
  LAMA | 13 |  | 15
  LABA: number analyzed (Participants) | 1 | 0 | 0
  LABA | 0 |  |
  LABA/LAMA: number analyzed (Participants) | 108 | 11 | 26
  LABA/LAMA | 36 | 11 | 26
  ICS/LABA: number analyzed (Participants) | 136 | 12 | 92
  ICS/LABA | 46 | 12 | 92
  Triple therapy (ICS/LABA/LAMA, SITT): number analyzed (Participants) | 134 | 7 | 97
  Triple therapy (ICS/LABA/LAMA, SITT) | 52 | 7 | 97
  MITT: number analyzed (Participants) | 49 | 4 | 50
  MITT | 22 | 4 | 50
  Theophylline: number analyzed (Participants) | 105 | 7 | 326
  Theophylline | 45 | 7 | 326
  MITT or SITT: number analyzed (Participants) | 183 | 11 | 147
  MITT or SITT | 74 | 11 | 147
  N-acetyl cysteine/carbocysteine: number analyzed (Participants) | 73 | 6 | 174
  N-acetyl cysteine/carbocysteine | 27 | 6 | 174

7. Secondary Outcome: Number of Participants With COPD Medication History
Description: Number of participants with COPD medication history were reported for following categories; Use the maintenance treatment, LAMA, LABA, LABA/LAMA, ICS/LABA, Triple therapy (ICS/LABA/LAMA, SITT), MITT, Theophylline, MITT or SITT, N-acetyl cysteine/carbocysteine. The measurement at Baseline visit (Day 1) was defined as Baseline. Participants may have received more than one COPD maintenance treatment. Hence, they may have counted in more than one category, so the total may not match to Number analyzed (N).
Time Frame: At Pre-Baseline (Within 1 month before Baseline [Day 1] visit)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Participants Presenting With Stable Disease | Cohort 2: Participants Presenting With a Moderate Acute Exacerbation Not Requiring Hospitalization | Cohort 3: Participants Requiring Hospitalization for an Acute Exacerbation
Number analyzed (Participants) | 797 | 71 | 615
Participants
  Use the maintenance treatment | 523 | 38 | 476
  LAMA | 75 | 0 | 15
  LABA | 1 | 0 | 0
  LABA/LAMA | 108 | 11 | 26
  ICS/LABA | 136 | 12 | 92
  Triple therapy (ICS/LABA/LAMA, SITT) | 134 | 7 | 98
  MITT | 49 | 4 | 50
  Theophylline | 105 | 7 | 330
  MITT or SITT | 183 | 11 | 148
  N-acetyl cysteine/carbocysteine | 73 | 6 | 175

8. Secondary Outcome: Chronic Obstructive Pulmonary Disease (COPD) Assessment Test (CAT) Scores by Historic Treatments at Indicated Time Point
Description: The CAT is an 8-item unidimensional measure of health status impairment in participants with COPD. Participants are scored on eight items (cough, phlegm, chest tightness, breathlessness, activity limitation, confidence, sleep and energy) on a scale of 0 (no impact) to 5 (worst possible impact) depending on their impact. The sum of scores for each item gives the participant's impact score ranging from 0 (no impact) to 40 (worst possible impact). Higher score indicates worst possible impact. CAT score by historic treatments including LAMA, LABA, LABA/LAMA, ICS/LABA, Triple therapy (ICS/LABA/LAMA, SITT), MITT, Theophylline, MITT or SITT, N-acetyl cysteine/carbocysteine were reported. Participants may have received more than one COPD maintenance treatment. Hence, they may have counted in more than one category, so the total may not match to Number analyzed (N). Mean and standard deviation (SD) values of CAT score assessments at 3 months are reported.
Time Frame: At 3 months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Cohort 1: Participants Presenting With Stable Disease | Cohort 2: Participants Presenting With a Moderate Acute Exacerbation Not Requiring Hospitalization | Cohort 3: Participants Requiring Hospitalization for an Acute Exacerbation
Number analyzed (Participants) | 797 | 71 | 615
Scores on a scale
  LAMA: number analyzed (Participants) | 75 | 0 | 15
  LAMA | 12.4 (8.27) |  | 19.5 (6.73)
  LABA: number analyzed (Participants) | 1 | 0 | 0
  LABA | 27.0 (NA) — NA indicates standard deviation could not be calculated for a single participant. |  |
  LABA/LAMA: number analyzed (Participants) | 107 | 11 | 26
  LABA/LAMA | 13.1 (9.03) | 16.8 (8.06) | 18.7 (6.54)
  ICS/LABA: number analyzed (Participants) | 136 | 12 | 92
  ICS/LABA | 14.8 (8.78) | 14.3 (5.07) | 18.0 (8.43)
  Triple therapy (ICS/LABA/LAMA, SITT): number analyzed (Participants) | 134 | 7 | 98
  Triple therapy (ICS/LABA/LAMA, SITT) | 13.7 (7.96) | 14.4 (8.04) | 21.5 (8.12)
  MITT: number analyzed (Participants) | 49 | 4 | 50
  MITT | 13.7 (9.15) | 15.8 (6.02) | 20.6 (7.49)
  Theophylline: number analyzed (Participants) | 105 | 7 | 330
  Theophylline | 14.1 (9.04) | 11.6 (6.32) | 19.4 (8.30)
  MITT or SITT: number analyzed (Participants) | 183 | 11 | 148
  MITT or SITT | 13.7 (8.27) | 14.9 (7.08) | 21.2 (7.90)
  N-acetyl cysteine/carbocysteine: number analyzed (Participants) | 73 | 6 | 175
  N-acetyl cysteine/carbocysteine | 13.1 (8.68) | 14.3 (9.54) | 19.3 (8.60)

9. Secondary Outcome: Modified Medical Research Council (mMRC) Score by Historic Treatments at Indicated Time Point
Description: The mMRC questionnaire predicts future mortality risk with mMRC. Participants are required to rate their disability due to shortness of breath on the 5-point mMRC scale ranging from 0 (no impact) to 4 (worst possible impact). Higher score indicates worst possible impact. The mMRC score by historic treatments including LAMA, LABA, LABA/LAMA, ICS/LABA, Triple therapy (ICS/LABA/LAMA, SITT), MITT, Theophylline, MITT or SITT, N-acetyl cysteine/carbocysteine were reported. Participants may have received more than one COPD maintenance treatment. Hence, they may have counted in more than one category, so the total may not match to Number analyzed (N). Mean and SD values of mMRC score assessments at 3 months are reported.
Time Frame: At 3 months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Cohort 1: Participants Presenting With Stable Disease | Cohort 2: Participants Presenting With a Moderate Acute Exacerbation Not Requiring Hospitalization | Cohort 3: Participants Requiring Hospitalization for an Acute Exacerbation
Number analyzed (Participants) | 797 | 71 | 615
Scores on a scale
  LAMA: number analyzed (Participants) | 75 | 0 | 15
  LAMA | 1.2 (0.91) |  | 2.1 (0.92)
  LABA: number analyzed (Participants) | 1 | 0 | 0
  LABA | 2.0 (NA) — NA indicates standard deviation could not be calculated for a single participant. |  |
  LABA/LAMA: number analyzed (Participants) | 107 | 11 | 26
  LABA/LAMA | 1.4 (1.02) | 1.8 (0.98) | 2.0 (1.17)
  ICS/LABA: number analyzed (Participants) | 136 | 12 | 92
  ICS/LABA | 1.7 (0.97) | 1.2 (1.19) | 2.1 (1.08)
  Triple therapy (ICS/LABA/LAMA, SITT): number analyzed (Participants) | 134 | 7 | 98
  Triple therapy (ICS/LABA/LAMA, SITT) | 1.7 (1.02) | 1.9 (0.69) | 2.4 (1.03)
  MITT: number analyzed (Participants) | 49 | 4 | 50
  MITT | 1.8 (1.03) | 2.3 (0.96) | 2.4 (1.09)
  Theophylline: number analyzed (Participants) | 105 | 7 | 330
  Theophylline | 1.7 (0.99) | 1.7 (0.95) | 2.2 (1.08)
  MITT or SITT: number analyzed (Participants) | 183 | 11 | 148
  MITT or SITT | 1.7 (1.03) | 2.0 (0.77) | 2.4 (1.04)
  N-acetyl cysteine/carbocysteine: number analyzed (Participants) | 73 | 6 | 175
  N-acetyl cysteine/carbocysteine | 1.7 (0.99) | 2.3 (1.03) | 1.9 (1.14)

10. Secondary Outcome: Number of Participants Requiring Hospitalization by Their Each Dyspnea, Eosinopenia, Consolidation, Acidemia and Atrial Fibrillation (DECAF) Risk Group
Description: DECAF is a 7-point scale with a minimum score of 0 (better outcome) and a maximum score of 6 (worse outcome). Higher score indicates worst outcome. It is used for assessment of severity of COPD exacerbation measures Dyspnea, Eosinopenia, consolidation, acidemia and atrial fibrillation. Number of participants requiring hospitalization by their each DECAF risk groups Mild (0-1 score), moderate (2 score), severe (3-6 score) were summarized. Participants who did not provide scores were categorized under "Missing". The measurement at Baseline visit (Day 1) was defined as Baseline.
Time Frame: Baseline (Day 1)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Participants Requiring Hospitalization for an Acute Exacerbation
Number analyzed (Participants) | 615
Participants
  Mild | 503
  Moderate | 49
  Severe | 5
  Missing | 58

11. Secondary Outcome: Number of Participants With at Least One Co-morbidity
Description: Number of participants with at least one co-morbidity were reported. Co-morbidities included Vascular disorders, Cardiac disorders, Respiratory, thoracic and mediastinal disorders, Metabolism and nutrition disorders, Infections and infestations, Gastrointestinal disorders, Reproductive system and breast disorders, Hepatobiliary disorders, Nervous system disorders, Renal and urinary disorders, Musculoskeletal and connective tissue disorders, Injury, poisoning and procedural complications, Psychiatric disorders, Endocrine disorders, Blood and lymphatic system disorders, Neoplasms benign, malignant and unspecified (including cysts and polyps), Skin and subcutaneous tissue disorders, Eye disorders, Investigations, General disorders and administration site conditions, Ear and labyrinth disorders, Congenital, familial and genetic disorders, Immune system disorders and Surgical and medical procedures).
Time Frame: Up to 3 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Participants Presenting With Stable Disease | Cohort 2: Participants Presenting With a Moderate Acute Exacerbation Not Requiring Hospitalization | Cohort 3: Participants Requiring Hospitalization for an Acute Exacerbation
Number analyzed (Participants) | 797 | 71 | 615
Participants | 512 | 52 | 571

12. Secondary Outcome: Number of Participants by Their Socio-economic Characteristics
Description: Questions were asked to participants to understand their following socio-economic factors associated with different patterns of COPD maintenance treatment;Education(No formal education, Elementary,Middle,High school-including vocational school, Bachelor's degree and above, Missing), Local permanent resident(No,Yes, Missing), Marriage condition(Married,Divorced/Separated,Widowed,Unmarried and Missing), With whom usually live(Live alone, With spouse, With one specific child, Take turns in different children's homes, Other relatives, Missing), National basic medical insurance (Insu.)(None,Government medical insu.,Urban employee medical insu., Urban resident medical insu., New cooperative medical insu., Urban and rural resident basic medical insu., Serious illness insu., Missing) and Commercial insu.(Yes,No,Missing). Participants may have provided more than one answers to questions. Hence, they may have counted in more than one category, so the total may not match to Number analyzed (N).
Time Frame: Baseline (Day 1)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Participants Presenting With Stable Disease | Cohort 2: Participants Presenting With a Moderate Acute Exacerbation Not Requiring Hospitalization | Cohort 3: Participants Requiring Hospitalization for an Acute Exacerbation
Number analyzed (Participants) | 797 | 71 | 615
Participants
  Education; No formal education | 38 | 1 | 40
  Education; Elementary school | 219 | 27 | 187
  Education; Middle school | 286 | 24 | 214
  Education; High school-including vocational school | 167 | 15 | 118
  Education; Bachelor's degree and above | 85 | 4 | 48
  Education; Missing | 2 | 0 | 8
  Local permanent resident; No | 69 | 7 | 89
  Local permanent resident; Yes | 726 | 64 | 518
  Local permanent resident; Missing | 2 | 0 | 8
  Marriage condition; Married | 717 | 66 | 516
  Marriage condition; Divorced/Separated | 19 | 2 | 14
  Marriage condition; Widowed | 54 | 3 | 71
  Marriage condition; Unmarried | 5 | 0 | 6
  Marriage condition; Missing | 2 | 0 | 8
  With whom usually live; Live alone | 84 | 7 | 64
  With whom usually live; With spouse | 612 | 53 | 415
  With whom usually live; With one specific child | 175 | 21 | 173
  With whom usually live; Take turns in different children's homes | 5 | 0 | 9
  With whom usually live; Other relatives | 7 | 0 | 0
  With whom usually live; Missing | 2 | 0 | 8
  National basic medical insurance; None | 9 | 1 | 3
  National basic medical insurance; Government medical insurance | 13 | 2 | 14
  National basic medical insurance; Urban employee medical insurance | 395 | 28 | 260
  National basic medical insurance; Urban resident medical insurance | 111 | 10 | 99
  National basic medical insurance; New cooperative medical insurance | 176 | 11 | 195
  National basic medical insurance; Urban and rural resident basic medical insurance | 89 | 19 | 31
  National basic medical insurance; Serious illness insurance | 2 | 0 | 2
  National basic medical insurance; Missing | 2 | 0 | 11
  Commercial insurance; No | 727 | 65 | 564
  Commercial insurance; Yes | 68 | 6 | 42
  Commercial insurance; Missing | 2 | 0 | 9

13. Secondary Outcome: Number of Participants by Their COPD Assessment Test (CAT) Scores at Indicated Time Points
Description: The CAT is an 8-item unidimensional measure of health status impairment in participants with COPD. Participants are scored on eight items (cough, phlegm, chest tightness, breathlessness, activity limitation, confidence, sleep and energy) on a scale of 0 (no impact) to 5 (worst possible impact) depending on their impact. The sum of scores for each item gives the participant's impact score ranging from 0 (no impact) to 40 (worst possible impact). Higher score indicates worst possible impact. Number of participants by their CAT scores were reported (<=10, 11 to 20, 21 to 30, 31 to 40). Participants who did not provide scores were categorized under "Missing". The measurement at Baseline visit (Day 1) was defined as Baseline.
Time Frame: Baseline (Day 1), Week 1, Discharge follow-up (up to 28 days) and at 3 months
Population: Analysis data set which included all participants from enrolled population excluding those who did not enter the study as they did not meet Protocol-defined eligibility criteria. Only those participants who were measured and analyzed (i.e., contributed data reported in the table) were included in the 'Overall Number of Participants Analyzed' field. 'Number Analyzed' signifies participants evaluable for the specified time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Participants Presenting With Stable Disease | Cohort 2: Participants Presenting With a Moderate Acute Exacerbation Not Requiring Hospitalization | Cohort 3: Participants Requiring Hospitalization for an Acute Exacerbation
Number analyzed (Participants) | 797 | 71 | 615
Participants
  Baseline (Day 1); Score <=10 | 300 | 20 | 109
  Baseline (Day 1); Scores 11 to 20 | 318 | 32 | 250
  Baseline (Day 1); Scores 21 to 30 | 148 | 18 | 199
  Baseline (Day 1); Scores 31 to 40 | 30 | 1 | 52
  Baseline (Day 1); Missing | 1 | 0 | 5
  Week 1; Score <=10: number analyzed (Participants) | 0 | 71 | 0
  Week 1; Score <=10 |  | 31 |
  Week 1; Scores 11 to 20: number analyzed (Participants) | 0 | 71 | 0
  Week 1; Scores 11 to 20 |  | 24 |
  Week 1; Scores 21 to 30: number analyzed (Participants) | 0 | 71 | 0
  Week 1; Scores 21 to 30 |  | 12 |
  Week 1; Scores 31 to 40: number analyzed (Participants) | 0 | 71 | 0
  Week 1; Scores 31 to 40 |  | 1 |
  Week 1; Missing: number analyzed (Participants) | 0 | 71 | 0
  Week 1; Missing |  | 3 |
  Discharge follow-up (up to 28 days); Score <=10: number analyzed (Participants) | 0 | 0 | 615
  Discharge follow-up (up to 28 days); Score <=10 |  |  | 229
  Discharge follow-up (up to 28 days); Scores 11 to 20: number analyzed (Participants) | 0 | 0 | 615
  Discharge follow-up (up to 28 days); Scores 11 to 20 |  |  | 246
  Discharge follow-up (up to 28 days); Scores 21 to 30: number analyzed (Participants) | 0 | 0 | 615
  Discharge follow-up (up to 28 days); Scores 21 to 30 |  |  | 95
  Discharge follow-up (up to 28 days); Scores 31 to 40: number analyzed (Participants) | 0 | 0 | 615
  Discharge follow-up (up to 28 days); Scores 31 to 40 |  |  | 19
  Discharge follow-up (up to 28 days); Missing: number analyzed (Participants) | 0 | 0 | 615
  Discharge follow-up (up to 28 days); Missing |  |  | 26
  At 3 months; Score <=10 | 420 | 38 | 239
  At 3 months; Score 11 to 20 | 238 | 21 | 213
  At 3 months; Score 21 to 30 | 90 | 7 | 71
  At 3 months; Score 31 to 40 | 21 | 1 | 22
  At 3 months; Missing | 28 | 4 | 70

14. Secondary Outcome: Number of Participants by Their Modified British Medical Research Council (mMRC) Score at Baseline
Description: The mMRC questionnaire predicts future mortality risk with mMRC. Participants are required to rate their disability due to shortness of breath on the 5-point mMRC scale ranging from 0 (no impact) to 4 (worst possible impact). Higher score indicates worst possible impact. Number of participants by their mMRC scores (Scores 0, 1, 2, 3 and 4) were summarized. Participants who did not provide scores were categorized under "Missing". The measurement at Baseline visit (Day 1) was defined as Baseline.
Time Frame: At Baseline (Day 1)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Participants Presenting With Stable Disease | Cohort 2: Participants Presenting With a Moderate Acute Exacerbation Not Requiring Hospitalization | Cohort 3: Participants Requiring Hospitalization for an Acute Exacerbation
Number analyzed (Participants) | 797 | 71 | 615
Participants
  Score 0 | 127 | 14 | 37
  Score 1 | 279 | 17 | 130
  Score 2 | 258 | 24 | 202
  Score 3 | 118 | 13 | 163
  Score 4 | 14 | 3 | 78
  Missing | 1 | 0 | 5

15. Secondary Outcome: Number of Participants Whose Prescribed Maintenance Treatment Was Stepped up, Stepped Down, Stopped, Switched, Remained the Same
Description: Number of participants whose prescribed maintenance therapy was stepped up (adding another maintenance therapy), stepped down (withdraw any of the maintenance medication but kept the maintenance therapy), stopped (stop all maintenance therapy), switched (between LAMA/LABA and ICS/LABA) or remained the same were reported. Participants whose treatment was not categorized in any of the above, were reported under Missing.
Time Frame: Up to 3 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Participants Presenting With Stable Disease | Cohort 2: Participants Presenting With a Moderate Acute Exacerbation Not Requiring Hospitalization | Cohort 3: Participants Requiring Hospitalization for an Acute Exacerbation
Number analyzed (Participants) | 797 | 71 | 615
Participants
  Stepped up | 67 | 4 | 180
  Stepped down | 26 | 1 | 14
  Stopped | 25 | 1 | 18
  Switched | 9 | 1 | 0
  Remained the same | 568 | 30 | 186
  Missing | 102 | 34 | 217

16. Secondary Outcome: Number of Participants Receiving COPD Maintenance Treatment at 3 Months
Description: Number of participants receiving COPD maintenance treatment including LAMA, LABA/LAMA, ICS/LABA, Triple therapy (ICS/LABA/LAMA, SITT), MITT, Theophylline, MITT or SITT, N-acetyl cysteine/carbocysteine were reported. Participants may have received more than one COPD maintenance treatment. Hence, they may have counted in more than one category, so the total may not match to Number analyzed (N).
Time Frame: At 3 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Participants Presenting With Stable Disease | Cohort 2: Participants Presenting With a Moderate Acute Exacerbation Not Requiring Hospitalization | Cohort 3: Participants Requiring Hospitalization for an Acute Exacerbation
Number analyzed (Participants) | 797 | 71 | 615
Participants
  LAMA | 92 | 6 | 20
  LABA/LAMA | 127 | 12 | 35
  ICS/LABA | 136 | 21 | 109
  Triple therapy (ICS/LABA/LAMA, SITT) | 240 | 11 | 181
  MITT | 51 | 4 | 46
  Theophylline | 93 | 6 | 82
  MITT or SITT | 291 | 15 | 227
  N-acetyl cysteine/carbocysteine | 80 | 7 | 52

ADVERSE EVENTS:
Time Frame: All-cause mortality, serious adverse events (SAEs) and non-serious adverse events (Non-SAEs) were collected up to 3 months
Description: All-cause mortality, SAEs and Non-SAEs were reported for Analysis Data Set (1483) since 24 participants from Enrolled Population (1507) did not enter the study as they did not meet Protocol-defined eligibility criteria. Analysis data set included all participants from enrolled population excluding those who did not enter the study as they did not meet Protocol-defined eligibility criteria.
Arm/Group | Cohort 1: Participants Presenting With Stable Disease | Cohort 2: Participants Presenting With a Moderate Acute Exacerbation Not Requiring Hospitalization | Cohort 3: Participants Requiring Hospitalization for an Acute Exacerbation
All-Cause Mortality (participants affected / at risk) | 4/797 | 0/71 | 2/615
Serious Adverse Events (participants affected / at risk) | 5/797 | 1/71 | 4/615
Other Adverse Events (participants affected / at risk) | 2/797 | 0/71 | 0/615
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Participants Presenting With Stable Disease (N=797) | Cohort 2: Participants Presenting With a Moderate Acute Exacerbation Not Requiring Hospitalization (N=71) | Cohort 3: Participants Requiring Hospitalization for an Acute Exacerbation (N=615)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 2
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0
Death (General disorders) | 0 | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Participants Presenting With Stable Disease (N=797) | Cohort 2: Participants Presenting With a Moderate Acute Exacerbation Not Requiring Hospitalization (N=71) | Cohort 3: Participants Requiring Hospitalization for an Acute Exacerbation (N=615)
Cataract (Eye disorders) | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-05-26): https://cdn.clinicaltrials.gov/large-docs/38/NCT04853238/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-14): https://cdn.clinicaltrials.gov/large-docs/38/NCT04853238/SAP_001.pdf